CLINICAL TRIAL: NCT00437944
Title: Relation Between Polymorphism in Genes Related to Kidney Disease and Renal Manifistations in Fabry Disease
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Other Study IDs: 50/06
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Fabry; Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The rational of the study is to try to predict which of the patients who suffer from Fabry disease will have End Stage Renal Disease. We hope to find correlation between certain modifier genes, previously related to renal disease, to renal disease in Fabry.

ELIGIBILITY:
Inclusion Criteria:Fabry disease -

Exclusion Criteria:none

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-05; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Gheona Altresko, Study Director